CLINICAL TRIAL: NCT02350257
Title: Internet-Based CBT for Children With Anxiety Disorders: Implementation in Clinical Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Eva Serlachius, Associate professor, child psychiatrist, MD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BIPSY RCT
Record Dates: First submitted 2015-01-19; First posted 2015-01-29 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Anxiety Disorders
Keywords: cognitive behavior therapy; child; randomized controlled trial; internet
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ICBT (Experimental): Internet-based cognitive behavior therapy
  Interventions: Behavioral: Internet-based CBT
- Supportive control (No Intervention): Control participants has weekly contact with a therapist and receives internet-based training in child directed play. Participants are informed that this training will not likely reduce anxiety.

INTERVENTIONS:
Behavioral: Internet-based CBT — 12 weeks of internet-based CBT
  Arms: ICBT

SUMMARY:
The primary objective of this study is to test the effectiveness of internet-delivered and therapist-guided internet-based cognitive behavior therapy (ICBT) for children with anxiety disorders (including social anxiety disorder, separation anxiety disorder, generalized anxiety disorder, panic disorder and specific phobia) in a randomized trial where participants will be allocated to either ICBT or to a supportive control condition. Non-responders (defined as those participants who still uphold their primary anxiety disorder after the ICBT treatment) will be offered traditional (face-to-face) CBT. Follow-ups are conducted at 3 and 12 months after treatment completion.

ELIGIBILITY:
Inclusion Criteria:

* A primary diagnosis of any of the following anxiety disorders, as defined by DSM-V (social anxiety disorder, separation anxiety disorder, generalized anxiety disorder, panic disorder or specific phobia)
* Age between 8 and 12 years
* Ability to read and write Swedish
* Daily access to the internet
* A parent that is able to co-participate in the treatment
* Participants on psychotropic medication must have been on a stable dose for the last 6 weeks prior to baseline assessment

Exclusion Criteria:

* Diagnosed with autism spectrum disorder, psychosis, bipolar disorder or severe eating disorder
* Present risk of suicide
* Ongoing substance dependence
* Completed CBT for any anxiety disorder within the last 6 months (defined as at least 5 sessions of CBT including in vivo exposure sessions)

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 131 (Actual)
Dates: Start 2015-03; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Clinician Severity Rating (CSR) | Baseline, 12 weeks after treatment starts, 3 and 12 months after treatment has ended
  Change from Baseline of anxiety disorder severity, after 12 weeks and at 3- and 12 months after treatment

SECONDARY OUTCOMES:
Presence of DSM Anxiety disorder | Assessed at Pre, Post, 3-month and 12-month Follow-up
Children´s Globas Assessment Scale (CGAS) | Assessed at Pre, Post, 3-month and 12-month Follow-up
Clinical Global Impression - Improvement (CGI-I) | Assessed at Post, 3-month and 12-month Follow-up
Revised Children´s Anxiety and Depression Scale - Child version (RCADS-C) | Assessed at Pre, Mid-3 weeks, Mid-6 weeks, Mid-9 weeks, Post, 3-month and 12-month Follow-up
Revised Children´s Anxiety and Depression Scale - Parent version (RCADS-P) | Assessed at Pre, Mid-3 weeks, Mid-6 weeks, Mid-9 weeks, Post, 3-month and 12-month Follow-up
KIDSCREEN-10 Child version | Assessed at Pre, Post, 3-month and 12-month Follow-up
  Quality of life
KIDSCREEN-10 Parent version | Assessed at Pre, Post, 3-month and 12-month Follow-up
  Quality of life
Education, Work and Social Adjustment Scale - Child version (EWSAS-C) | Assessed at Pre, Mid-6 weeks, Post, 3-month and 12-month Follow-up
Education, Work and Social Adjustment Scale - Parent version (EWSAS-P) | Assessed at Pre, Mid-6 weeks, Post, 3-month and 12-month Follow-up
Hospital Anxiety and Depression Scale - Parents (HADS) | Assessed at Pre
Technology Acceptance Scale - Child (TAS-C) | Assessed at Mid-3 weeks and Post
  Perceived usefulness and perceived ease of use
Technology Acceptance Scale - Parent (TAS-P) | Assessed at Mid-3 weeks and Post
  Perceived usefulness and perceived ease of use
Trimbos/iMTA questionnaire for Costs associated with Psychiatric Illness (TIC-P) | Assessed at Pre, Post, 3-month and 12-month Follow-up
Measurement of compliance to exposure assignments and anxiety levels, through mobile app | During the 12 weeks of ICBT
  Participants register anxiety levels in adjunction to exposure exercises, with a smartphone app
Unintended treatment effects | Assessed at Post
Specific Phobia Questionnaire - Child version (SPQ-C) | Assessed at Pre, Mid-3 weeks, Mid-6 weeks, Mid-9 weeks, Post, 3-month and 12-month Follow-up
Specific Phobia Questionnaire - Parent version (SPQ-P) | Assessed at Pre, Mid-3 weeks, Mid-6 weeks, Mid-9 weeks, Post, 3-month and 12-month Follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- BUP CPF, Stockholm, Sweden

REFERENCES:
- [Derived] Jolstedt M, Wahlund T, Lenhard F, Ljotsson B, Mataix-Cols D, Nord M, Ost LG, Hogstrom J, Serlachius E, Vigerland S. Efficacy and cost-effectiveness of therapist-guided internet cognitive behavioural therapy for paediatric anxiety disorders: a single-centre, single-blind, randomised controlled trial. Lancet Child Adolesc Health. 2018 Nov;2(11):792-801. doi: 10.1016/S2352-4642(18)30275-X. Epub 2018 Sep 18. PMID 30241993
- See also: Barninternetprojektet — http://www.bup.se/bip